CLINICAL TRIAL: NCT05117125
Title: Biomarkers for Prediction of and Diagnosis of Ventilator-associated Pneumonia
Brief Title: Biomarkers for Ventilator-associated Pneumonia
Acronym: VAPmarkers
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00219
Record Dates: First submitted 2021-10-15; First posted 2021-11-11 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mini-BAL Plasma Protected specimen brushes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- VAP: Enrolled participants that fully meet the criteria of VAP.
  Interventions: Diagnostic Test: Heparin-binding protein; Diagnostic Test: Interleukin-26; Diagnostic Test: Microbiome; Diagnostic Test: Bacterial transcriptome; Diagnostic Test: Proteome
- Suspect VAP: Enrolled participants that develop signs of VAP but lack some variable, for instace new radiographic infiltrate or microbiological finding compatible with VAP.
  Interventions: Diagnostic Test: Heparin-binding protein; Diagnostic Test: Interleukin-26; Diagnostic Test: Microbiome; Diagnostic Test: Proteome
- No VAP: Enrolled participants that do not develop VAP.
  Interventions: Diagnostic Test: Heparin-binding protein; Diagnostic Test: Interleukin-26; Diagnostic Test: Microbiome; Diagnostic Test: Proteome

INTERVENTIONS:
Diagnostic Test: Heparin-binding protein — Evaluation of the specificity and sensitivity of HBP as diagnostic biomarker for VAP.
  Other Names: HBP
Diagnostic Test: Interleukin-26 — Evaluation of the specificity and sensitivity of IL-26 as diagnostic biomarker for VAP.
  Other Names: IL-26
Diagnostic Test: Microbiome — Evaluation of the specificity and sensitivity of the lung microbiome as prognostic biomarker for VAP.
Diagnostic Test: Bacterial transcriptome — Evaluation of the specificity and sensitivity of the bacterial transcriptome as prognostic biomarker for treatment failure of VAP.
  Groups: VAP
Diagnostic Test: Proteome — Evaluation of the specificity and sensitivity of the proteome in mini-BAL as biomarker for VAP.

SUMMARY:
The purpose of this study is to evaluate different peptide biomarkers, variations in the microbiome and patterns in the bacterial transcriptome as prognostic or diagnostic biomarkers of VAP.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an intensive care unit
* Intubation within last 24 hours
* Anticipated mechanical ventilation of at least 48 hours

Exclusion Criteria:

* FiO2 above 70% or PEEP above 15
* Severe coagulopathy (spontaneous PK(INR) >1.8 or thrombocytes <50). Prophylaxis treatment dose of LMWH or factor Xa inhibitors/NOAC is not an exclusion criteria. If higher doses of these substances are administered, the responsible clinician should be consulted before sample collection.
* Ongoing infection of the lungs at admission to the ICU.
* Severely elevated or instable intracranial pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General intensive care unit population.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HBP concentration over time | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Change in concentration (ng/ml) compared to baseline.
Change in IL-26 over time | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Change in concentration (ng/ml) compared to baseline.
HBP at VAP diagnosis | VAP day 1 compared to No VAP day 3
  Concentration at VAP day 1, compared to day 3 in patients with no VAP. ROC curves, specificity and sensitivity as diagnostic biomarker.
IL-26 at VAP diagnosis | VAP day 1 compared to No VAP day 3
  Concentration at VAP day 1, compared to day 3 in patients with no VAP. ROC curves, specificity and sensitivity as diagnostic biomarker.

SECONDARY OUTCOMES:
Diversity of microbiome | Day 1 and 3, and VAP day 1.
  Changes in alpha and beta diversity as prognostic biomarker for VAP. Cases that develop VAP are compared to cases with no VAP.
Bacterial transcriptome patterns | VAP day 1
  Patterns in the bacterial gene expression that predict antibiotic drug treatment failure.

OTHER OUTCOMES:
Diagnostic certainty of VAP | At VAP day 1
  A scale from 0-100 of the diagnostic certainty by ICU physicians and nurses
Change in CRP concentration | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare cases with VAP to No VAP
Change in Differential blood cell counts | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare cases with VAP to No VAP
Change in PCT concentration | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare cases with VAP to No VAP
Change in lactate concentration | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare cases with VAP to No VAP
Routine bacterial culture results | When mini-BAL is collected
  Results from cultures at the clinical microbiology laboratory. Results will be correlated to bacterial species identification in mini-BAL.
Change in Acute Physiology And Chronic Health Evaluation II (APACHE II) | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare score between cases with VAP and no VAP.
Change in Sequential Organ Failure Assessment (SOFA) | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare score between cases with VAP and no VAP.
Change in Simplified Acute Physiology Score III (Saps3) | Day 1, 3 and in selected patients day 7 and 14. In patients with VAP also VAP day 1, 3 and 7.
  Compare score between cases with VAP and no VAP.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Paulsson, PhD MD, Principal Investigator — Skane University Hospital; Fredrik Sjövall, PhD MD, Study Chair — Skane University Hospital
Locations (5):
- Vestre Viken, Drammen, Norway
- Hospital de São Francisco Xavier, Lisbon, Portugal
- Sweden (3):
  - Skåne University Hospital, Dept. of Infectious diseases, Lund
  - Skåne university Hospital, ICU, Malmo
  - Karolinska University Hospital, ICU, Solna

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in published articles will be shared with investigators after deidentification upon request.
Supporting Information: Study Protocol
Time Frame: IPD will be available from 6 months to 5 years after publication.
Access Criteria: Approval of the relevant ethical board is necessary for access

REFERENCES:
- [Background] Paulsson M, Cardenas EI, Che KF, Brundin B, Smith M, Qvarfordt I, Linden A. TLR4-mediated release of heparin-binding protein in human airways: a co-stimulatory role for IL-26. Front Immunol. 2023 May 10;14:1178135. doi: 10.3389/fimmu.2023.1178135. eCollection 2023. PMID 37234157
- [Background] Paulsson M, Thelaus L, Riesbeck K, Qvarfordt I, Smith ME, Linden A, Linder A. Heparin-binding protein in lower airway samples as a biomarker for pneumonia. Respir Res. 2021 Jun 8;22(1):174. doi: 10.1186/s12931-021-01764-2. PMID 34103069
- See also: Related Info — https://www.medicin.lu.se/forskning/patientstudier/vap-markorstudien